CLINICAL TRIAL: NCT02295306
Title: The Evaluation of a Respiratory Volume Monitor in Patients Undergoing Overnight Polysomnography
Brief Title: Overnight Polysomnography and Respiratory Volume Monitor
Status: Active, not recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Respiratory Motion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 10880
Record Dates: First submitted 2014-09-26; First posted 2014-11-20 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: OSA, polysomnography, ExSpiron monitor
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Respiratory Volume Monitor (RVM, ExSpiron) — Connecting patient to the ExSpiron monitor and continuous ExSpiron data collection during the patient's polysomnography (PSG)

SUMMARY:
Sleep disordered breathing; specifically obstructive sleep apnea (OSA) is a disease affecting 8-12% of the general population and often more than 70% of the bariatric surgical population. OSA is characterized by the repetitive collapse of the upper airway, causing a reduction or cessation in airflow and decreases in oxygen saturation. These events are resolved by arousals from sleep, reducing sleep quality and leading to excessive daytime sleepiness. An in-laboratory polysomnography (PSG) is the gold standard for the diagnosis of OSA.

Previous studies have established obstructive sleep apnea (OSA) as a potential independent risk factor for postoperative complications, adverse surgical outcomes, and longer hospital stays.

Patients with OSA have an increase in postoperative complications, the most frequent being oxygen desaturation, postoperative atelectasis and increased postoperative pain. Despite the clear risks, OSA remains under diagnosed with an estimated 25-30% of patients at a high risk for OSA. It has been suggested that OSA events may be even more frequent post operatively because of the residual effects of anesthesia and the use of potent pain medications such as opioids. Postoperatively apneas often go undetected and untreated. The use of supplemental O2 may mask any desaturations and there is no convenient technology to noninvasively monitor ventilation to detect apnea and hypopnea in post-surgical patients.

New advances in technology and digital signal processing have led to the development of an impedance based Respiratory Volume Monitor (RVM). The RVM (ExSpiron™, Respiratory Motion, Inc.; Waltham, MA) has been shown to provide accurate real-time, continuous, non-invasive measurements of tidal volume (TV), minute ventilation (MV) and respiratory rate (RR). Our main hypotheses are that the non-invasive, impedance-based RVM monitor will accurately reflect TV, RR and MV during sleep and will detect apneas and hypopneas accurately.

DETAILED DESCRIPTION:
This is an observational pilot study to evaluate the clinical applicability of the ExSpiron Respiratory Volume Monitor (RVM) in patients with suspected sleep apnea. Previous work has demonstrated the ability of the RVM to provide non-invasive, real-time, continuous measurements of respiratory parameters (MV, TV, and RR) but those studies have not specifically looked at patients during sleep or patients with sleep disordered breathing.

Previously there was no device capable of providing, continuous, non-invasive, real time measurements of ventilatory status such as minute ventilation, tidal volume and RR. The ExSpiron system utilizing impedance based technology and proprietary algorithms (Respiratory Motion Inc., Waltham, MA) have been developed to obtain these measurements.

Respiratory Motion, Inc. has previously evaluated ExSpiron measurements of respiratory parameters (MV, TV and RR) in studies of adult volunteer subjects. Stimulus leads delivered an alternating minimal current (1.5 mA) at a frequency of 50 kHz and recording leads recorded differential voltages to calculate impedance. Subject data (height, weight, age, gender, chest circumference) were measured. The studies showed that using the optimal lead placement configuration, algorithms based on chest wall impedance and respiratory pattern analysis provided provided RVM measurements and ExSpiron curves which correlated strongly with spirometry volumes and spirometry curves.

A large percentage of patients in the general surgical population have undiagnosed OSA. This population is at increased risk of adverse perioperative respiratory complications. Assessment and management of perioperative respiratory function and early intervention when indicated is a multifaceted, complex task often complicated by the unavailability of an accurate and continuous monitoring system that can demonstrate apnea and hypopnea to guide clinical decision making. The ExSpiron system is designed for these patients and is intended to address some of the limitations of the current generation of hospital monitors as listed below:

In the, non-ventilated patient, current monitoring devices do not provide objective non-invasive, continuous real time measurements of important respiratory parameters MV, TV and RR that reflect respiratory competence, nor do they provide adequate assessment of apnea and hypopnea.

Current monitoring of non-intubated patients mostly relies on oximetry data, subjective clinical assessment which measures respiration and not ventilation and rarely transcutaneous CO2 measurements. In appropriate clinical settings, the ExSpiron system can provide direct quantitative measure of ventilation (MV, TV and RR) that can be used in the detection of apnea and hypopnea.

Precise apnea and hypopnea assessment.

Most if not all of the gaps left by current respiratory assessment technologies may be filled by a non-invasive monitor such as the one proposed for use in this study. There are many potential applications for this technology including: use in peri-procedural environment to evaluate the effects of medication on ventilation and detection of apnea/hypopnea. In addition, it may be useful in clinical decision making regarding medication adjustments of pain management protocols, evaluation ventilatory status prior to extubation and evaluation of the need for reintubation, but also trending of respiratory patterns to avoid risky emergency airway management interventions.

New advances in technology and digital signal processing have led to the development of an impedance based Respiratory Volume Monitor (RVM). The RVM (ExSpiron™, Respiratory Motion, Inc.; Waltham, MA) has been shown to provide accurate real-time, continuous, non-invasive measurements of tidal volume (TV), minute ventilation (MV) and respiratory rate (RR). Our main hypotheses are that the non-invasive, impedance-based RVM monitor will accurately reflect TV, RR and MV during sleep and will detect apneas and hypopneas accurately.

Main Hypothesis: The ExSpiron monitor accurately reflects apnea and hypopnea events compared to standard polysomnography. The ExSpiron monitor is able to distinguish between central and obstructive apneic events.

Secondary Hypothesis: 1) Correlation of MV% as compared to % predicted with comorbidities (e.g. hypertension and metabolic syndrome), 2)Correlation of MV changes as compared to MV% predicted with oxygen desaturation index (ODI), 3) evaluation breathing patterns before and after obstruction, 4) evaluation of breathing patterns in different types of apnea (central, obstructive and mixed).

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients referred to the sleep lab for a polysomnography for suspicion of sleep disordered breathing aged ≥ 18 years. Ability to provide written informed consent.

Exclusion Criteria:

- Patients not competent to give informed consent, patients with implantable electronic devices, such as pacemakers, stimulators, etc. pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients referred to the sleep laboratory at Tufts Medical Center for a standard polysomnogram (PSG) are eligible to be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between number and duration of apnea events measured as AHI (apnea hypopnea index) assessed by standard polysomnography versus Exspiron monitor | Duration of polysomnography study, usually 1 overnight assessment

SECONDARY OUTCOMES:
Ability of the Exspiron monitor to distinguish between central and obstructive apnea events. There is no unit measurement for this comparison | Duration of polysomnography study, usually 1 overnight assessment

CONTACTS AND LOCATIONS:
Overall Officials: Roman Schumann, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States